CLINICAL TRIAL: NCT02710786
Title: Long-term Resolution of Comorbidites After Gastric Bypass
Brief Title: Comorbidity After Gastric Bypass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other); The Scandinavian Obesity Surgery Registry (Unknown)
Responsible Party: Sponsor
Other Study IDs: Comorb
Record Dates: First submitted 2016-02-18; First posted 2016-03-17 (Estimated); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Severe Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gastric bypass: Patients undergoing gastric bypass
  Interventions: Procedure: Gastric bypass

INTERVENTIONS:
Procedure: Gastric bypass — Gastric bypass surgery, i.e., small gastric pouch and excluded main stomach

SUMMARY:
To evaluate effect on comorbid disease and weight loss in the long-term (>five years) after Roux-en-Y gastric bypass (RYGB) surgery for severe obesity.

DETAILED DESCRIPTION:
Individuals with severe obesity frequently have comorbid diseases, e.g. diabetes, hypertension, hyperlipidemia, and sleep apnea. We will study the remission rate and weight loss in the long-term (10 years) after Roux-en-Y gastric bypass (RYGB) surgery in a nationwide large group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Registered individuals in Scandinavian Obesity Surgery Registry (SOReg) having had gastric bypass

Exclusion Criteria:

* All other operations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals undergoing gastric bypass
Sampling Method: Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2007-05 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in comorbid conditions, as defined by use of pharmacological treatment | 10 years
  Remission of diabetes mellitus, hypertension, dyslipidemia, and depression as defined by use of pharmacological treatment, and sleep apnea as defined by use of CPAP. Data will be collected from SOReg.

SECONDARY OUTCOMES:
Number of patients with pathological laboratory data (corresponding to the studied comorbid conditions) | 10 years
  Glucose, HbA1c, LDL, HDL, triglycerides, and blood pressure
Weight loss | 10 years
  Peroperative weight (in kg) minus current weight (in kg)
BMI loss | 10 years
  Peroperative BMI minus current BMI. Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Ingemar Näslund, Study Chair — Scandinavian Obesity Surgery Registry
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No